CLINICAL TRIAL: NCT07389629
Title: The Efficacy and Safety of Iparomlimab and Tuvonralimab (QL1706) Combined With Lenvatinib as Neoadjuvant Therapy in Renal Cancer With Partial Nephrectomy Indications But High Surgical Risk：A Single Arm, Phase II Clinical Study
Brief Title: Iparomlimab and Tuvonralimab (QL1706) Combination With Lenvatinib as Neoadjuvant Therapy for ccRCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, ZHOU FANGJIAN, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-FXY-071
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Iparomlimab and Tuvonralimab; Clear Cell Renal Cell Carcinoma; Neoadjuvant Therapy
Keywords: Iparomlimab and Tuvonralimab; Clear Cell Renal Cell Carcinoma; Neoadjuvant therapy
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Iparomlimab and Tuvonralimab (QL1706) combined with Lenvatinib as neoadjuvant therapy (Experimental): Lenvatinib Treatment Lenvatinib (8mg [body weight < 60 kg] or 12 mg [body weight ≥ 60 kg]) orally once daily, with or without food.
  Intravenous Infusion of QL1706(Injection) Infuse QL1706 at a dose of 5mg/kg intravenously every three weeks, constituting one treatment cycle, a total of 2 or 4 cycles.
  Interventions: Drug: QL1706 Combined With Lenvatinib

INTERVENTIONS:
Drug: QL1706 Combined With Lenvatinib — Lenvatinib Treatment Lenvatinib (8mg [body weight < 60 kg] or 12 mg [body weight ≥ 60 kg]) orally once daily, with or without food.
  Intravenous Infusion of QL1706(Injection) Infuse QL1706 at a dose of 5mg/kg intravenously every three weeks, constituting one treatment cycle, a total of 2 or 4 cycles.

SUMMARY:
Through the combination of aparolitovorelli monoclonal antibody and lenvatinib neoadjuvant therapy, partial nephrectomy can be successfully and safely performed in patients with localized renal cell carcinoma (T1N0M0 or T2N0M0) who have indications for kidney preservation surgery but have difficulty in preserving the kidney (R.E.N.A.L. score >= 10).

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign a written informed consent form (ICF).
2. Age at the time of enrollment is >= 18 and under 80 years old, with no gender restrictions.
3. The physical fitness score of the Eastern Cooperative Oncology Group (ECOG) in the United States is 0 or 1;
4. Expected survival period >= 3 months.
5. Preoperative biopsy pathology confirmed renal clear cell carcinoma or renal cell carcinoma mainly composed of clear cell carcinoma;
6. ECOG score 0 or 1;
7. The patient is willing to undergo kidney preservation surgery;
8. Indications for kidney preservation surgery are available, but limited renal cancer with high difficulty of kidney preservation surgery (stage T1N0M0 or T2N0M0, must meet R.E.N.A.L. score >= 10);
9. At least one measurable lesion (according to mRECIST v1.1 standard) that is suitable for repeated and accurate measurements.
10. Good organ function, screening laboratory test results meet the following criteria: (1) Hematology (no blood components or cell growth factors are allowed to support treatment within 2 weeks before starting treatment): a. Absolute neutrophil count (ANC) >= 1.5 × 10^9/L (1500/mm^3); b. Platelet count (PLT) >= 100 × 10^9/L (100000/mm^3); c. Hemoglobin (HB) >= 90 g/L; (2) Liver: a. Serum total bilirubin (TBIL) <= 1.5 × ULN; b. Alanine transaminase (ALT) and aspartate transaminase (AST) <= 2.5 × ULN; For subjects with liver metastases, AST and ALT are <= 5 × ULN, while serum albumin (ALB) is >= 28g/L. Coagulation function: international normalized ratio (INR) and activated partial thromboplastin time (APTT) are <= 1.5 × ULN;
11. The subjects are willing and able to comply with the scheduled visits, treatment plans, laboratory tests, and other requirements of the study.

Exclusion Criteria:

1. lymph node metastasis;
2. The tumor surrounds the renal artery;
3. Renal vein cancer thrombus;
4. Diffuse tumor growth, with no clear boundary from normal renal parenchyma;
5. General poor condition, anesthesia assessment cannot tolerate general anesthesia surgery;
6. Have serious cardiovascular and cerebrovascular diseases, uncontrollable hypertension and diabetes;
7. Patients who have long-term use of immunosuppressants after organ transplantation;
8. Patients who are currently using immunosuppressive drugs;
9. Patients with clear infection or fever;
10. Patients with T-cell lymphoma and myeloma;
11. Patients who have concurrent malignant tumors, are currently undergoing treatment for other benign or malignant tumors, or have a history of other malignant tumors within the past six months;
12. Metastatic renal cell carcinoma.
13. Received Chinese herbal medicine or immunomodulatory drugs with anti-tumor indications within 14 days prior to the first use of the investigational drug;
14. Perform systematic treatment (including thymosin, interferon, interleukin, except for local use to control pleural effusion).
15. Suffering from active or potentially recurrent autoimmune diseases, except for vitiligo, hair loss, psoriasis, or eczema that do not require systemic treatment; Hypothyroidism caused by autoimmune thyroiditis only requires stable doses of hormone replacement therapy; Type I diabetes requiring only a stable dose of insulin replacement therapy.
16. Simultaneously enrolled in another clinical study, unless it is an observational, non interventional clinical study or a follow-up period of an interventional study.
17. Known history of mental illness, drug abuse, alcoholism, or drug use.
18. Pregnant or lactating women.
19. Any past or current illness, treatment, or laboratory test abnormalities may confuse the research results, affect the full participation of the subjects in the study, or participation in the study may not be in the best interests of the subjects.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-11-21 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Decline rate of tumor R.E.N.A.L score | Evaluation at the end of Cycle 2 or 4 (each cycle is 21 days) of QL1706 treatment

SECONDARY OUTCOMES:
ORR | Evaluation at the end of Cycle 2 or 4 (each cycle is 21 days) of QL1706 treatment
  Objective Response Rate (ORR) based on RECIST 1.1 criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No